CLINICAL TRIAL: NCT00660972
Title: First-Phase Viral Decay Rates in Treatment-Naive Subjects Initiating Treatment With Raltegravir (RAL) and Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF): A Pilot Study
Brief Title: Study of Viral Load Decay Rates in HIV Infected Participants Starting Treatment With Raltegravir (RAL) and Emtricitabine/Tenofovir Disoproxil Fumarate (TDF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Adult AIDS Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5248; 10532 (Registry Identifier: DAIDS ES); ACTG A5248
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Integrase Inhibitors; HIV Nucleoside Reverse Transcriptase Inhibitors; Treatment Naive; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

ARMS (1):
- 1 (Experimental): Oral RAL and FTC/TDF for 72 weeks
  Interventions: Drug: Raltegravir; Drug: Emtricitabine/tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Raltegravir — 400 mg tablet taken orally twice daily
  Other Names: RAL
Drug: Emtricitabine/tenofovir disoproxil fumarate — Fixed dose tablet containing 200 mg emtricitabine and 300 mg tenofovir disoproxil fumarate taken once daily. FTC/TDF will not be provided by the study and must be obtained by the particpant's health care provider.
  Other Names: FTC/TDF

SUMMARY:
The HIV integrase inhibitor, raltegravir (RAL), which was recently approved by the FDA, has been shown in several trials to be highly effective. The purpose of this trial is to estimate the viral load decay rate in treatment-naive HIV infected participants receiving RAL and emtricitabine/tenofovir disoproxil fumarate (FTC/TDF).

DETAILED DESCRIPTION:
Recent data suggests that early virologic response to HIV interventions may be predictive of long-term virologic outcomes. Defining early decay in viral load through carefully performed studies of viral dynamics may be a useful tool for assessing the likely outcome of long-term treatment. It may also be a useful screening tool to define which combinations should be studied further. In this trial, the viral load decay rate will be estimated in HIV infected, treatment-naive participants receiving RAL and FTC/TDF.

This study will last approximately 72 weeks. All participants will take RAL and FTC/TDF for 72 weeks. RAL will be provided by the study. FTC/TDF will not be provided.

This study will consist of 16 study visits. These visits will occur at study entry, Days 2, 7, 10, 14, 21, 28, and 56, and Weeks 12, 16, 20, 24, 36, 48, 60, and 72. Blood collection and pharmacokinetic studies will occur at all study visits. Self-reported adherence assessments will be submitted at each visit. A targeted physical exam will occur at most visits. Liver function tests and urine collection will occur at select visits. Pregnancy tests will occur whenever pregnancy is suspected.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Antiretroviral treatment naive
* Viral load at least 10,000 and less than 300,000 copies/ml within 42 days prior to study entry
* Agree to use appropriate form of contraception. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Received HIV-specific immunizations within 6 months prior to study entry
* Received immunizations within 6 months prior to study entry
* Known allergy or sensitivity to study drugs
* Any participant with an acute AIDS-defining opportunistic infection (OI) who is not clinically stable or who has not been on therapy for the OI for at least 30 days prior to study entry
* Treatment with immune modulators or any investigational therapy within 30 days prior to study entry
* Evidence of HIV seroconversion within 6 months prior to study entry
* Illness requiring systemic treatment and/or hospitalization
* Substance abuse that, in the opinion of the investigator, would interfere with adherence to study requirements
* Requirement for any current medications that are prohibited with any study medication. More information on this criterion can be found in the protocol.
* Evidence of any major resistance-associated mutation on any genotype performed prior to study entry or at the time of screening. More information on this criterion can be found in the protocol.
* Abnormal laboratory values. More information on this criterion can be found in the protocol.
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Viral load decay rates | Through Day 56

SECONDARY OUTCOMES:
Viral load decay rates | From Weeks 24 to 72
Proportion of participants with a viral load less than 50 copies/ml | At Weeks 24, 48, and 72
Safety and tolerability. More information on this criterion can be found in the protocol. | Throughout study
CD4 and CD8 count | Throughout study
Resistance mutations to RAL, FTC, and TDF | Throughout study
Minimum concentration (Cmin) for RAL, FTC, and TDF | Throughout study
Changes in viral load | At Day 7
Self-reported adherence | Throughout study
Cell-associated proviral DNA, LTR circular DNA, and integrated proviral DNA | Throughout study
Viral load | From Week 24 to Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Andrade, MD, MPH, Study Chair — Johns Hopkins University
Locations (15):
- United States (15):
  - UCSD Antiviral Research Center CRS, San Diego, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Brigham and Women's Hospital Therapeutics Clinical Research Site (BWH TCRS) CRS, Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - Harlem ACTG CRS, New York, New York
  - Trillium Health ACTG CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - MetroHealth CRS, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Houston AIDS Research Team CRS, Houston, Texas

REFERENCES:
- [Background] Evering TH, Markowitz M. Raltegravir: an integrase inhibitor for HIV-1. Expert Opin Investig Drugs. 2008 Mar;17(3):413-22. doi: 10.1517/13543784.17.3.413. PMID 18321239
- [Background] Sedaghat AR, Dinoso JB, Shen L, Wilke CO, Siliciano RF. Decay dynamics of HIV-1 depend on the inhibited stages of the viral life cycle. Proc Natl Acad Sci U S A. 2008 Mar 25;105(12):4832-7. doi: 10.1073/pnas.0711372105. Epub 2008 Mar 24. PMID 18362342
- [Derived] Funderburg NT, Xu D, Playford MP, Joshi AA, Andrade A, Kuritzkes DR, Lederman MM, Mehta NN. Treatment of HIV infection with a raltegravir-based regimen increases LDL levels, but improves HDL cholesterol efflux capacity. Antivir Ther. 2017;22(1):71-75. doi: 10.3851/IMP3091. Epub 2016 Oct 14. PMID 27740536
- [Derived] Funderburg NT, Andrade A, Chan ES, Rosenkranz SL, Lu D, Clagett B, Pilch-Cooper HA, Rodriguez B, Feinberg J, Daar E, Mellors J, Kuritzkes D, Jacobson JM, Lederman MM. Dynamics of immune reconstitution and activation markers in HIV+ treatment-naive patients treated with raltegravir, tenofovir disoproxil fumarate and emtricitabine. PLoS One. 2013 Dec 18;8(12):e83514. doi: 10.1371/journal.pone.0083514. eCollection 2013. PMID 24367599